CLINICAL TRIAL: NCT02130947
Title: Randomized, Controlled Study of an Exercise Intervention Program for Patients With Metastatic Castration-Resistant Prostate Cancer Receiving Either Abiraterone or Enzalutamide
Brief Title: Exercise Intervention for Pts With Metastatic Castration-Resistant Prostate Cancer Receiving Abiraterone or Enzalutamide
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: We were not able to accrue any participants.
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: LCCC 1339; 14-0177 (Other: UNC IRB)
Record Dates: First submitted 2014-05-01; First posted 2014-05-06 (Estimated); Last update posted 2016-02-11 (Estimated); Status verified 2016-02

CONDITIONS: Metastatic Castration Resistant Prostate Cancer (mCRPC)
Keywords: Metastatic Castration Resistant Prostate Cancer; Prostate Cancer; mCRPC; Pilot Study; UNC Lineberger; Exercise
MeSH Terms: conditions — Prostatic Neoplasms; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise Intervention Arm (Experimental): The exercise intervention will consist of a combination of aerobic (cardiovascular exercise) and strength training (emphasis of the intervention) 3 times per week for 12 weeks with each session lasting ~1.5 hours.
  Interventions: Behavioral: Exercise
- Non-Exercise Control Arm (No Intervention): Participants in the Non-Exercise Control Arm will not exercise for 12 weeks.

INTERVENTIONS:
Behavioral: Exercise
  Arms: Exercise Intervention Arm

SUMMARY:
This randomized pilot study will be conducted in men with metastatic castration resistant prostate cancer (mCRPC) within 3 months of initiating abiraterone or enzalutamide. The purpose of this pilot study is to evaluate the effects of a 12 week exercise intervention in mCRPC patients who have recently started on additional androgen suppression therapy.

DETAILED DESCRIPTION:
This randomized pilot study will be conducted in men with metastatic castration resistant prostate cancer (mCRPC) within 3 months of initiating abiraterone or enzalutamide. The purpose of this pilot study is to evaluate the effects of a 12 week exercise intervention in mCRPC patients who have recently started on additional androgen suppression therapy. The investigators will also explore the effects of the exercise training on biomarkers of inflammation-hormonal status and their potential association with changes in lean mass and function.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years of age
2. Metastatic disease that has progressed despite castrate levels of testosterone (surgically or medically castrated, with testosterone levels of < 50 ng/dL)
3. No prior chemotherapy
4. Initiated therapy with either abiraterone plus a glucocorticoid or enzalutamide within the 3 months prior to randomization
5. Ability to engage safely in moderate exercise as determined by their treating physician
6. Not previously engaged in regular exercise training (>1-2 d/wk for > 30 min/d) in the past 6 months
7. Be able to speak and read English

Exclusion Criteria:

1. Any condition that causes severe pain with exertion
2. History of bone fractures
3. Active cardiovascular disease including any of the following:

   * New York Heart Association (NYHA) Grade II or greater congestive heart failure
   * History of myocardial infarction or unstable angina within 6 months prior to Day 1
   * History of stroke or transient ischemic attack within 6 months prior to Day 1
4. Acute or chronic respiratory disease
5. Acute or chronic bone/joint/muscular abnormalities compromising their ability to exercise
6. Neurological conditions that affect balance and, or muscle strength
7. Dementia, altered mental status or any psychiatric condition prohibiting the understanding or rendering of informed consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-04; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Change in lean mass between mCPRC patients undergoing a 12-week exercise intervention (intervention group) and mCPRC patients who do not undergo the exercise intervention (control group) | 12 weeks
  DEXA (Dual-energy X-ray absorptiometry) scans will measure lean mass at baseline and after the 12-week intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony C Hackney, Ph.D., D.Sc., Principal Investigator — University of North Carolina
Locations (1):
- Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina, United States

REFERENCES:
- See also: Lineberger Comprehensive Cancer Center website — http://unclineberger.org/
- See also: National Cancer Institute (NCI) website — http://www.cancer.gov/